CLINICAL TRIAL: NCT00974155
Title: Randomised Clinical Trial Comparing Early Medication Change (EMC) Strategy With Treatment as Usual (TAU) in Patients With Major Depressive Disorder - the EMC Trial
Brief Title: The Early Medication Change (EMC) Trial
Acronym: EMC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: K. Lieb (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor-Investigator, K. Lieb, Study Principal Investigator, Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-016; 2008-008280-96 (EudraCT Number)
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Depression
Keywords: Major; Depression; Disorder
MeSH Terms: conditions — Depression; Disease | interventions — Escitalopram; Venlafaxine Hydrochloride; Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EMC (Early Medication Change) (Experimental)
  Interventions: Drug: Escitalopram, venlafaxine, lithium
- TAU (Therapy As Usual) (Active Comparator)
  Interventions: Drug: Escitalopram, venlafaxine

INTERVENTIONS:
Drug: Escitalopram, venlafaxine, lithium — oral application, highest tolerable dose, once daily
  Arms: EMC (Early Medication Change)
Drug: Escitalopram, venlafaxine — oral application, highest tolerable dose, once daily
  Arms: TAU (Therapy As Usual)

SUMMARY:
The EMC trial investigates for the first time prospectively whether Major Depression Disorder patients with non-improvement after 14 days of antidepressive treatment with EMC are more likely to become remitters compared to patients treated according to current guidelines, i.e., with a medication change after 28 days of treatment in case of non-response.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder (MDD), first episode or recurrent, according to DSM-IV
* HAMD17 score of ≥18 pts.
* Age between 18 and 65 years and age ≤ 60 years at the time of the first depressive episode
* Ability of subject to understand character and individual consequences of clinical trial
* Signed and dated informed consent of the subject must be available before start of any specific trial procedures.

Exclusion Criteria:

* Acute risk of suicide needing an intervention not comprised by protocol treatment (e.g. electroconvulsive therapy)
* Patients with a lifetime DSM-IV diagnosis of dementia, schizophrenia, schizoaffective disorder, bipolar disorder
* Patients with a current DSM-IV diagnosis of posttraumatic stress disorder, obsessive-compulsive disorder, anxiety disorder, or eating disorder and the requirement of a treatment not comprised by protocol treatment
* Patients with DSM-IV substance dependency requiring acute detoxification
* Depression due to organic brain disorder, e.g. Multiple Sclerosis and Parkinson's Disease
* Women who are pregnant, breastfeeding or planning to become pregnant during the trial
* Women who are not sterile by surgery or for more than two years postmenopausal or women with childbearing potential who not practicing a medically accepted contraception during trial
* Patients currently taking antidepressant medication, which has been started within the 2-4 weeks prior to study begin and a continuation of this antidepressant medication is clinically indicated
* A clear history of non-response to an adequate treatment trial in the current major depressive episode to any protocol antidepressant. A "clear history of non-response" has to be assumed, when the following criteria are fulfilled:

  * ad Escitalopram: Treatment with a mDDD ≥ 15 mg/d for 4 weeks or CPL 15-80 ng/ml for four weeks without response, i.e. a symptom reduction ≥ 50% between start and end of treatment.
  * ad Venlafaxine: Treatment with a mDDD ≥ 300 mg/d for 4 weeks or CPL 195-400 ng/ml for four weeks without response, i.e. a symptom reduction ≥ 50% between start and end of treatment;
  * ad Lithium: Treatment with CPL 0.6-0.8 mmol Li+ for four weeks without response, i.e. a symptom reduction ≥ 50% between start and end of treatment
* History of medical or psychological condition, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or render the patient at high risk from treatment complications
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product
* Clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation. Such conditions may include gastrointestinal, cardiovascular, vascular disease, pulmonary/respiratory, hepatic impairment, renal, metabolic diseases, endocrinological, neurological, immune-deficiency, hematopoietic disease, or malignancies as determined by medical history, physical examination, or laboratory tests
* Participation in other clinical trials during the present clinical trial or within the last 6 months
* Medical or psychological condition that would not permit signing of informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 889 (Actual)
Dates: Start 2009-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Remission from MDD on day 56, defined as a HAMD17 sum score ≤ 7, in non-improvers on day 14 (n=192) | 8 weeks

SECONDARY OUTCOMES:
Response, defined as a HAMD17 sum score decrease ≥50% on day 56 | 8 weeks
Absolute change of HAMD17 sum score | 8 weeks
Remission defined as IDS score ≤ 11 on day 56 | 8 weeks
Response defined as IDS score decrease ≥50% on day 56 | 8 weeks
Absolute change in SF12 subscales "physical component score" and "mental component score" | 8 weeks
Remission from MDD, defined as a HAMD17 sum score ≤ 7 on day 56 (subgroups of improvers on day 14) | 8 weeks
Time to remission and time to response according to IDS and HAMD17 | 8 weeks
Occurrence of adverse events, UKU ratings at all visits, relevant laboratory data and deviations from normal ECG | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Lieb, Prof., Principal Investigator — Clinic of Psychiatry and Psychotherapy Mainz
Locations (1):
- University Medical Center of the Johannes Gutenberg-University, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Derived] Engelmann J, Murck H, Wagner S, Zillich L, Streit F, Herzog DP, Braus DF, Tadic A, Lieb K, Muller MB. Routinely accessible parameters of mineralocorticoid receptor function, depression subtypes and response prediction: a post-hoc analysis from the early medication change trial in major depressive disorder. World J Biol Psychiatry. 2022 Oct;23(8):631-642. doi: 10.1080/15622975.2021.2020334. Epub 2022 Jan 25. PMID 34985381
- [Derived] Engelmann J, Wagner S, Solheid A, Herzog DP, Dreimuller N, Muller MB, Tadic A, Hiemke C, Lieb K. Tolerability of High-Dose Venlafaxine After Switch From Escitalopram in Nonresponding Patients With Major Depressive Disorder. J Clin Psychopharmacol. 2021 Jan/Feb 01;41(1):62-66. doi: 10.1097/JCP.0000000000001312. PMID 33208708
- [Derived] Dreimuller N, Lieb K, Tadic A, Engelmann J, Wollschlager D, Wagner S. Body mass index (BMI) in major depressive disorder and its effects on depressive symptomatology and antidepressant response. J Affect Disord. 2019 Sep 1;256:524-531. doi: 10.1016/j.jad.2019.06.067. Epub 2019 Jul 2. PMID 31280076
- [Derived] Engelmann J, Wagner S, Wollschlager D, Kaaden S, Schlicht KF, Dreimuller N, Braus DF, Muller MB, Tuscher O, Frieling H, Tadic A, Lieb K. Higher BDNF plasma levels are associated with a normalization of memory dysfunctions during an antidepressant treatment. Eur Arch Psychiatry Clin Neurosci. 2020 Mar;270(2):183-193. doi: 10.1007/s00406-019-01006-z. Epub 2019 Mar 30. PMID 30929060
- [Derived] Dreimuller N, Wagner S, Engel A, Braus DF, Roll SC, Elsner S, Tadic A, Lieb K. Predictors of the effectiveness of an early medication change strategy in patients with major depressive disorder. BMC Psychiatry. 2019 Jan 14;19(1):24. doi: 10.1186/s12888-019-2014-x. PMID 30642308
- [Derived] Lieb K, Dreimuller N, Wagner S, Schlicht K, Falter T, Neyazi A, Muller-Engling L, Bleich S, Tadic A, Frieling H. BDNF Plasma Levels and BDNF Exon IV Promoter Methylation as Predictors for Antidepressant Treatment Response. Front Psychiatry. 2018 Oct 26;9:511. doi: 10.3389/fpsyt.2018.00511. eCollection 2018. PMID 30459647
- [Derived] Wagner S, Helmreich I, Wollschlager D, Meyer K, Kaaden S, Reiff J, Roll SC, Braus D, Tuscher O, Muller-Dahlhaus F, Tadic A, Lieb K. Early improvement of executive test performance during antidepressant treatment predicts treatment outcome in patients with Major Depressive Disorder. PLoS One. 2018 Apr 18;13(4):e0194574. doi: 10.1371/journal.pone.0194574. eCollection 2018. PMID 29668746
- [Derived] Wagner S, Kayser S, Engelmann J, Schlicht KF, Dreimuller N, Tuscher O, Muller-Dahlhaus F, Braus DF, Tadic A, Neyazi A, Frieling H, Lieb K. Plasma brain-derived neurotrophic factor (pBDNF) and executive dysfunctions in patients with major depressive disorder. World J Biol Psychiatry. 2019 Sep;20(7):519-530. doi: 10.1080/15622975.2018.1425478. Epub 2018 Feb 2. PMID 29334322
- [Derived] Herzog DP, Wagner S, Ruckes C, Tadic A, Roll SC, Harter M, Lieb K. Guideline adherence of antidepressant treatment in outpatients with major depressive disorder: a naturalistic study. Eur Arch Psychiatry Clin Neurosci. 2017 Dec;267(8):711-721. doi: 10.1007/s00406-017-0798-6. Epub 2017 Apr 18. PMID 28421334
- [Derived] Tadic A, Wagner S, Gorbulev S, Dahmen N, Hiemke C, Braus DF, Lieb K. Peripheral blood and neuropsychological markers for the onset of action of antidepressant drugs in patients with Major Depressive Disorder. BMC Psychiatry. 2011 Jan 26;11:16. doi: 10.1186/1471-244X-11-16. PMID 21269443
- [Derived] Tadic A, Gorbulev S, Dahmen N, Hiemke C, Braus DF, Roschke J, van Calker D, Wachtlin D, Kronfeld K, Gorbauch T, Seibert-Grafe M, Lieb K; EMC Study Group. Rationale and design of the randomised clinical trial comparing early medication change (EMC) strategy with treatment as usual (TAU) in patients with major depressive disorder--the EMC trial. Trials. 2010 Feb 26;11:21. doi: 10.1186/1745-6215-11-21. PMID 20187947